CLINICAL TRIAL: NCT00135343
Title: A Pilot Study of Atazanavir/Ritonavir/Efavirenz as a Nucleoside Sparing Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AI424-121
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2008-07

CONDITIONS: HIV Infections
Keywords: HIV/AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ritonavir; efavirenz; Atazanavir Sulfate

ARMS (2):
- A (Experimental)
  Interventions: Drug: Atazanvir/ritonavir + efavirenz
- B (Experimental)
  Interventions: Drug: Atazanvir/ritonavir + efavirenz

INTERVENTIONS:
Drug: Atazanvir/ritonavir + efavirenz — Capsules (ATV and RTV) Tablets (EFV), Oral, ATV 300 mg + RTV 100 mg + EFV 600 mg, Once daily, 48 weeks.
  Other Names: Reyataz & Sustiva
  Arms: A
Drug: Atazanvir/ritonavir + efavirenz — Capsules (ATV and RTV) Tablets (EFV), Oral ATV 400 mg + RTV 100 mg + EFV 600 mg, Once daily, 48 weeks.
  Other Names: Reyataz & Sustiva
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a novel nucleoside sparing regimen containing atazanavir, ritonavir and efavirenz, using two different doses of atazanavir.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* HIV positive with plasma HIV RNA viral load of ≥ 1000 copies/mL and CD4 cell count of ≥ 50 cells/mm3
* Antiretroviral (ARV) naive prior to enrollment
* Normal plasma triglycerides ≤ 200 mg/dL
* Women of child-bearing age must use effective barrier contraception

Exclusion Criteria:

* Pregnancy or breast feeding
* Evidence of resistance to antiretroviral drugs
* History of elevated blood cholesterol or triglycerides
* History of diabetes
* Hypersensitivity to any component of the study drugs
* Any cholesterol or triglyceride lowering medications in the past six months
* Use of growth hormone, megestrol acetate, or anabolic steroids in the past six months
* Imprisonment or involuntary incarceration for medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10

PRIMARY OUTCOMES:
Mean percent change from baseline in fasting plasma triglycerides at Week 8

SECONDARY OUTCOMES:
Incidence of grade 2-4 elevation of fasting plasma triglycerides at Week (Wk) 8, 24 and 48
The mean percent change from baseline in fasting plasma triglycerides at Wk 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (15):
  - Local Institution, San Francisco, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Atlantis, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, South Miami, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Boston, Massachusetts
  - Local Institution, Berkley, Michigan
  - Local Institution, St Louis, Missouri
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Clumbia, South Carolina
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Hampton, Virginia